CLINICAL TRIAL: NCT02742246
Title: Efficacy and Mechanisms of Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) for Alcohol Use Disorders
Brief Title: Efficacy and Mechanisms of CBT4CBT for Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1511016759; 1R01AA024122-01A1 (NIH); 1K02AA027300-01A1 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-04-18 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment as usual (TAU) (No Intervention): This is the regular treatment a participant would normally receive at the clinic and generally includes individual and/or group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks and include issues such as teaching about the treatment program, teaching important ideas about recovery, increasing knowledge about specific problems participants may have with addiction and/or demonstrating new ways of coping with skills designed to fit their lifestyle. Participants will also be asked to complete a brief questionnaire and to provide urine and breath specimens for alcohol and drug testing once each week.
- Individual clinician-provided CBT (Active Comparator): This is individual treatment provided by a trained Cognitive Behavioral Therapy (CBT) clinician who will focus on teaching skills to understand and change participants behaviors to help them avoid alcohol use. Sessions with the clinician will generally last for 1 hour one time per week for 8 weeks. Participants will also be asked to complete a brief questionnaire and to provide urine and breath specimens for alcohol and drug testing once each week.
  Interventions: Behavioral: Individual clinician-provided CBT
- CBT4CBT (Experimental): In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on. The CBT4CBT program will cover the same skills as the individual clinician-provided CBT, only here it will be done by a computer. Participants will be taught how to use the computer program by a staff member and will be asked to spend about 8 hours using the program (approximately one hour per week) at the clinic.Participants will also be asked to complete a brief questionnaire and to provide urine and breath specimens for alcohol and drug testing once each week.
  Interventions: Behavioral: CBT4CBT

INTERVENTIONS:
Behavioral: Individual clinician-provided CBT — Individual clinician-provided CBT
  Arms: Individual clinician-provided CBT
Behavioral: CBT4CBT — CBT computer program assisted therapy
  Arms: CBT4CBT

SUMMARY:
Evaluate the efficacy of CBT4CBT and clinician-delivered CBT relative to standard treatment for reducing alcohol use

DETAILED DESCRIPTION:
Evaluate the efficacy of Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) and clinician-delivered Cognitive Behavioral Therapy (CBT) relative to standard treatment for reducing alcohol use through an 8-week randomized trial with 6-month follow-up. Our primary hypothesis is that either form of CBT will be more effective than standard treatment at increasing the percentage of days abstinent during treatment (8 weeks) and through the follow-up (6 months), assessed via Timeline FollowBack interviews.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be included who:

* Are 18 years of age or older.
* Are applying for outpatient alcohol treatment and meet current DSM-5 criteria for alcohol use disorder, consuming at least 14/7 drinks (men/women) per week with at least 4 heavy drinking days reported in the past 28 days,
* Are sufficiently stable for 8 weeks of outpatient treatment and can commit to a 6-month follow-up
* Are willing to provide locator information for follow-up, and
* Are fluent in English and have a 6th grade or higher reading level.

Exclusion Criteria:

Individuals will be excluded who:

* Have an untreated bipolar or schizophrenic disorder,
* Have a current legal case pending such that incarceration during the 8-week protocol is likely,
* Have been prescribed an alcohol pharmacotherapy (e.g., disulfiram, naltrexone) within the past two weeks, or
* Are physically dependent on alcohol, opioids or benzodiazepines such that immediate medical detoxification is necessary for safety purposes (individuals demonstrating significant withdrawal symptoms would be eligible for re-screening following brief medical detoxification, which is arranged by RCS staff at triage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kiluk, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - MCCA, Bridgeport, Connecticut
  - SATU, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiluk BD, Benitez B, DeVito EE, Frankforter TL, LaPaglia DM, O'Malley SS, Nich C. A Digital Cognitive Behavioral Therapy Program for Adults With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2435205. doi: 10.1001/jamanetworkopen.2024.35205. PMID 39325452

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initiated is the number that attended at least 1 treatment session. Every attempt was made to get post treatment and follow up interviews on everyone randomized, regardless of how much of the active treatment the participant received.
Groups:
- Individual Clinician-provided Cognitive Behavioral Therapy (CBT): This is individual treatment provided by a trained Cognitive Behavioral Therapy (CBT) clinician who will focus on teaching skills to understand and change participants behaviors to help them avoid alcohol use. Sessions with the clinician will generally last for 1 hour one time per week for 8 weeks. Participants will also be asked to complete a brief questionnaire and to provide urine and breath specimens for alcohol and drug testing once each week.
  Individual clinician-provided CBT: Individual clinician-provided CBT
- Computer Based Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT): In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on. The CBT4CBT program will cover the same skills as the individual clinician-provided CBT, only here it will be done by a computer. Participants will be taught how to use the computer program by a staff member and will be asked to spend about 8 hours using the program (approximately one hour per week) at the clinic.Participants will also be asked to complete a brief questionnaire and to provide urine and breath specimens for alcohol and drug testing once each week.
  CBT4CBT: CBT computer program assisted therapy
Period: Overall Study
Arm/Group | Standard Treatment as Usual (TAU) | Individual Clinician-provided Cognitive Behavioral Therapy (CBT) | Computer Based Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT)
Started (Number randomized to treatment assignment) | 34 | 32 | 33
Completed | 21 | 16 | 22
Not Completed | 13 | 16 | 11
Not completed — Never initiated treatment | 5 | 3 | 1
Not completed — dropped out during treatment | 7 | 13 | 10
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized to a treatment Assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment as Usual (TAU) | Individual Clinician-provided CBT | CBT4CBT | Total
Number analyzed (Participants) | 34 | 32 | 33 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14) | 45.3 (12.6) | 46.8 (11.6) | 45.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 14 | 33
  Male | 22 | 25 | 19 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 9 | 3 | 7 | 19
  Ethnicity: Minority | 22 | 16 | 18 | 56
  Ethnicity: Unknkown | 3 | 13 | 8 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 13 | 17 | 17 | 47
  Race: African-American | 16 | 13 | 10 | 39
  Race: Marked Hispanic only | 3 | 1 | 4 | 8
  Race: Multiracial | 1 | 1 | 1 | 3
  Race: Other | 0 | 0 | 1 | 1
  Race: Unknown | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 33 | 99
Completed High School [Count of Participants; unit: Participants] | 32 | 31 | 27 | 90
never married/living alone [Count of Participants; unit: Participants] | 27 | 24 | 25 | 76
Unemployed [Count of Participants; unit: Participants] | 21 | 17 | 21 | 59
Lifetime anxiety disorder [Count of Participants; unit: Participants] | 3 | 4 | 8 | 15
Lifetime major depression [Count of Participants; unit: Participants] | 7 | 12 | 10 | 29
AUD Severity Rating [Count of Participants; unit: Participants] — Alcohol Use Disorder (AUD) Severity Rating is a standardized scale from the Structured Clinical Interview Diagnosis (SCID) that assess Alcohol Use Disorder based on the DSM -V criteria. The scale ranges from (0-3 ) 0= absent, 1=Mild, 2 = Moderate, 3 = Severe
  Participants
    Mild | 3 | 1 | 1 | 5
    Moderate | 8 | 7 | 7 | 22
    Severe | 23 | 24 | 25 | 72
Audit Score 16 or higher [Count of Participants; unit: Participants] — The Alcohol Use Disorders Identification Test (AUDIT) is a 10 item questionnaire. The Range of the score is (0 - 40) with higher scores meaning more severe alcohol use disorder. The cut off score of 16 was used to create a dichotomous variable with the value of 0 = No, (AUDIT score less than 16) and 1= Yes,( AUDIT Score is 16 or higher)
  Participants | 25 | 24 | 28 | 77
On probation/ court referred [Count of Participants; unit: Participants] | 16 | 11 | 7 | 34
Mean days of alcohol use during the past 28 days [Mean (Standard Deviation); unit: days] | 14.2 (7.8) | 12.8 (8.6) | 14.5 (9.2) | 13.8 (8.5)
Mean days of heavy drinking during the past 28 days [Mean (Standard Deviation); unit: days] — Heavy drinking is considered 4 or more drinks for a women in a 24 hour period and 5 or more drinks for men in a 24 hour period
  days | 8.9 (8.1) | 9.1 (8.4) | 10.8 (9) | 9.6 (8.5)
Mean number of Drinks per drinking day during the past 28 days [Mean (Standard Deviation); unit: drinks per drinking day] — The average number of drinks a person consumed on a day that they drank alcohol
  drinks per drinking day | 6.3 (4) | 7.1 (4) | 8.7 (8) | 7.4 (5.7)
Mean number of Years of regular alcohol use [Mean (Standard Deviation); unit: years] — number of years of alcohol use where the frequency was 3 or more times per week
  years | 20.1 (13.8) | 22 (13.2) | 18.8 (12.7) | 20.3 (13.2)
Audit Score [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a 10 item questionnaire. The Range of the total score is (0 - 40) with higher scores meaning more severe alcohol use disorder.
  units on a scale | 20.7 (9) | 21.4 (8.6) | 23.9 (6.3) | 22 (8.1)
pre-treatment SCID Alcohol Symptom Count [Mean (Standard Deviation); unit: symptoms] | 7.1 (2.7) | 7.8 (2.4) | 8.6 (2.9) | 7.8 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Abstinent From Alcohol Use During Treatment as Measured by Timeline Follow Back
Description: The Timeline Follow Back is a calendar-based questionnaire used to assess alcohol use-consumption variables and can be used to measure alcohol use over time. This outcome was updated upon results entry. Presented are the percent days abstinent from alcohol use.
Time Frame: Baseline up to 8 weeks
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Standard Treatment as Usual (TAU) | Individual Clinician-provided CBT | CBT4CBT
Number analyzed (Participants) | 34 | 32 | 33
percentage of days abstinent
  Baseline | 49.26 (27.84) | 53.73 (29.80) | 47.57 (31.82)
  Week 4: number analyzed (Participants) | 31 | 31 | 30
  Week 4 | 63.25 (29.81) | 69.93 (29.42) | 71.07 (28.24)
  Week 8: number analyzed (Participants) | 28 | 29 | 29
  Week 8 | 69.26 (26.18) | 68.10 (29.85) | 75.12 (25.08)
Statistical Analysis 1: Comparison: Standard Treatment as Usual (TAU) vs Individual Clinician-provided CBT vs CBT4CBT; Test type: Superiority; p = 0.11, Regression, Linear — Group by Time interaction

2. Primary Outcome: Percentage of Days Abstinent From Alcohol Use During 6-month Follow-up Period as Measured by Timeline Follow Back
Description: The Timeline Follow Back is a calendar-based questionnaire used to assess alcohol use-consumption variables and can be used to measure change over time. This outcome was updated upon results entry. Presented are the percent days abstinent from alcohol use summarized monthly.
Time Frame: from end of treatment at week 8 up to 6 months
Population: Intention to treat process was used for data collection. All randomized participants were tracked and follow up data collection was attempted for the 6 months post treatment. Contact attempts were at 1 month, 3 month and 6 month post treatment. Analysis population numbers start at the number of randomized participants that completed the 1 month post treatment interview. Months 2 and 3 numbers reflex number of randomized participants that attended the 3 month post treatment interview and so on.
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Standard Treatment as Usual (TAU) | Individual Clinician-provided CBT | CBT4CBT
Number analyzed (Participants) | 28 | 29 | 27
percentage of days abstinent
  End of Treatment | 69.26 (26.18) | 68.10 (29.85) | 73.28 (25.03)
  Follow Up Month 1 | 66.71 (32.06) | 75.86 (29.29) | 74.74 (32.64)
  Follow Up Month 2: number analyzed (Participants) | 25 | 27 | 26
  Follow Up Month 2 | 63.86 (35.61) | 71.96 (30.91) | 77.06 (28.59)
  Follow Up Month 3: number analyzed (Participants) | 25 | 27 | 26
  Follow Up Month 3 | 55.14 (37.53) | 68.12 (33.15) | 82.55 (22.84)
  Follow Up Month 4: number analyzed (Participants) | 23 | 26 | 24
  Follow Up Month 4 | 67.70 (36.48) | 63.74 (35.90) | 82.14 (23.07)
  Follow Up Month 5: number analyzed (Participants) | 23 | 26 | 24
  Follow Up Month 5 | 68.17 (37.16) | 68.27 (37.13) | 85.12 (23.66)
  Follow Up Month 6: number analyzed (Participants) | 23 | 26 | 24
  Follow Up Month 6 | 69.57 (34.39) | 70.19 (35.11) | 82.59 (25.26)
Statistical Analysis 1: Comparison: Standard Treatment as Usual (TAU) vs Individual Clinician-provided CBT vs CBT4CBT; Test type: Superiority; p = 0.14, Regression, Linear — Group by time interaction

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | Standard Treatment as Usual (TAU) | Individual Clinician-provided CBT | CBT4CBT
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 8/34 | 1/32 | 7/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment as Usual (TAU) (N=34) | Individual Clinician-provided CBT (N=32) | CBT4CBT (N=33)
Hospitalization for Alcohol Use symptoms (Psychiatric disorders) | 2 (5) | 0 (0) | 2 (2)
Hospitalization for Detox (Psychiatric disorders) | 4 (4) | 0 (0) | 2 (3)
Hospitalization for Mental health (Psychiatric disorders) | 1 (1) | 1 (2) | 1 (1)
Hospitalization for Lacerations to body (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hospitalization for Intestinal issue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02742246/Prot_SAP_000.pdf